CLINICAL TRIAL: NCT06179615
Title: Surface Hardness and Wear Resistance of Prefabricated and CAD/CAM Milled Artificial Teeth: A Cross-over Clinical Study
Brief Title: Surface Hardness and Wear Characteristics of Prefabricated and CAD/CAM Milled Artificial Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Aisha Zakaria Hashem Mostafa, Professor of prosthodontics, Mansoura University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A11080622
Record Dates: First submitted 2023-12-11; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Surface Hardness and Wear Resistance of Artificial Teeth

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- complete denture with prefabricated artificial teeth (Other): complete denture constructed with prefabricated artificial teeth and inserted in the patient mouth to be used for 3, 6 months
  Interventions: Other: surface hardness test for denture teeth; Other: wear resistance of denture teeth measurement
- complete denture with CAD\CAM milled artificial teeth (Other): complete denture constructed with CAD\CAM Milled artificial teeth and inserted in the patient mouth to be used for 3, 6 months
  Interventions: Other: surface hardness test for denture teeth; Other: wear resistance of denture teeth measurement

INTERVENTIONS:
Other: surface hardness test for denture teeth — surface hardness test of denture teeth at insertion then after 6 months of use
Other: wear resistance of denture teeth measurement — 2D, Vertical wear, 3D Volumetric wear were measured for denture teeth

SUMMARY:
Purpose: This study aimed to assess the 3-dimentional wear )3D) (volumetric loss) and 2-dimentional wear (2D) (vertical loss) and surface hardness of ready-made (prefabricated) and CAD/CAM milled artificial denture teeth.

material and methods: In a cross-over study design, ten completely edentulous patients were randomly chosen for this study and given two complete dentures. The first complete denture was constructed with pre-fabricated teeth. The second complete denture was constructed with CAD\CAM milled teeth. The complete denture teeth were 3D scanned at the time of insertion (T0), after three months (T3), and after six months (T6) of denture insertion. Utilizing 3D surface superimposition techniques, the vertical (2D wear), and Volumatic (3D wear) material loss were measured. The hardness of the teeth were evaluated at the time of denture insertion (T0) then after 6 months (T6) of denture insertion by Vickers hardness test. Statistical analysis was done using SPSS software. Paired groups were compared by paired t test. Significant difference was considered if P ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* completely edentulous
* angle class I maxillomandibular relations

Exclusion Criteria:

* Angle's class II, III maxillomandibular relation
* systemic disease that affect the bone and soft tissue health

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
wear resistance of denture artificial teeth | 6 months after denture use
  2D, 3D wear of denture teeth were measured using denture scanning and superimposition of the sanning at insertion to that after 3, 6 months using Exocad soft ware
surface hardness of the denture artificial teeth | 6 months after denture use
  the measurement of surface hardness was done using Vickers's test. this measurements was done at insertion then after 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry, Mansoura univeristy, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abozaed HW, Ali SA, Mostafa AZ. Patient satisfaction and oral health-related quality of life for prefabricated teeth versus CAD-CAM milled acrylic resin denture teeth. A crossover clinical trial. BMC Oral Health. 2025 Oct 10;25(1):1601. doi: 10.1186/s12903-025-06834-1. PMID 41073957